CLINICAL TRIAL: NCT01390558
Title: Gait Parameters of Persons With Down Syndrome With and Without Orthotics Using GaitRite
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, David Oleson, Associate Professor, Oregon Health and Science University
Other Study IDs: Gait Parameters Down Syndrome
Record Dates: First submitted 2011-06-27; First posted 2011-07-11 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Orthotics; Gait Analysis
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Persons with Down Syndrome who use orthotics: Orthotic users
  Interventions: Procedure: custom orthotics
- Persons with Down Syndrome who do not use orthotics: Non orthotic users

INTERVENTIONS:
Procedure: custom orthotics — Orthotics are fabricated uniquely for each patient and use molds or casts of their foot as the template. They are fabricated by a licensed orthotist. There is no device or brand name other than custom orthotics.
  Groups: Persons with Down Syndrome who use orthotics

SUMMARY:
This is a research study of persons with Down Syndrome between 2 and 80 years old who are independently walking. The purpose of this study is to see what effect orthotics have on how people with Down Syndrome walk.

ELIGIBILITY:
Inclusion Criteria:

* Down Syndrome, independent walkers

Exclusion Criteria:

* Down Syndrome, not independently walking

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with Down Syndrome followed in Down Syndrome clinic Persons with Down Syndrome recruited in the community
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Gait will be measured with the GaitRite gait evaluation system. | 3 years
  Specific temporal and spatial parameters of gait will be measured with the GaitRite gait evaluation system. Subjects will walk with and without their orthotics. Measurement will be by changes in the previously noted gait parameters between the orthotics and non-orthotics groups.

SECONDARY OUTCOMES:
Elucidate patterns in the development of walking in persons with Down Syndrome using GaitRite®. | 3 years
  The previously described parameters of gait as measured by the GaitRite system will be used to establish an overview of the development of gait in persons with Down Syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Child Development and Rehabilitation Center, Portland, Oregon, United States